CLINICAL TRIAL: NCT01758146
Title: Impact of Obesity on the Efficacy of Endocrine Therapy With Aromatase Inhibitors in Postmenopausal Patients With Early Breast Cancer
Brief Title: Impact of Obesity on the Efficacy of Endocrine Therapy With Aromatase Inhibitors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMI
Record Dates: First submitted 2012-12-01; First posted 2013-01-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; obesity; aromatase inhibitors; postmenopausal
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Tamoxifen; Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A- Letrozole (Experimental): Aromatase inhibitor- letrozole 2.5mg once daily for 5 years
  Interventions: Drug: Letrozole
- Arm B- Tamoxifen (Active Comparator): Tamoxifen 20 mg once daily for 5 years
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — 20 mg once daily for 5 years
  Other Names: Canditam, Nolvadex
  Arms: Arm B- Tamoxifen
Drug: Letrozole — Letroz, Femara, Letronat
  Other Names: 2.5 mg once daily for 5 years
  Arms: Arm A- Letrozole

SUMMARY:
To see the impact of obesity on the efficacy of adjuvant endocrine therapy with aromatase inhibitors in postmenopausal patients with early breast cancer in terms of:

i) Locoregional recurrence ii) Distant metastases iii) Disease-free survival iv) Overall survival

DETAILED DESCRIPTION:
The relationship between obesity and breast cancer is a complex one. Obesity is a risk factor for the development of breast cancer in postmenopausal women and has been linked to an increased risk of recurrence and decreased survival as compared to patients with normal weight.

The hypothesis that led to this study is that the amount of total-body aromatization capacity indicated by body mass index (BMI). In postmenopausal women and in premenopausal women with ovarian suppression, the major source of serum estrogens is the fat tissue, in which precursors are metabolized to estrogens by the enzyme aromatase. Thus, an increase in BMI leads to an increase in total-body aromatization and, consequently, an increase in oestrogen serum levels, which impact on breast cancer. Taken together, this suggests that BMI may serve as a useful surrogate parameter for total-body aromatization and eventually may be a practicable tool to tailor aromatase inhibitors (AIs) therapy for individual patients.

The study will include 360, postmenopausal patients with early breast cancer who have hormones receptor positive tumour as defined by the expression of oestrogen receptor (ER) and/or progesterone receptor (PR). Patients will be randomly assigned to receive tamoxifen 20 mg once daily or AIs (letrozole 2.5mg/ anastrozole 1mg/exemestane 25mg) once daily for five years. Patients with a tumour stage IB, IC, or II irrespective of nodal stage (<10 positive nodes) will be included. Weight and height will be taken at baseline for calculation of BMI according to the WHO criteria. The frequency of adverse events will be used to assess safety throughout the study.

The primary end point will be disease-free survival (DFS). Secondary end points will be recurrence-free survival and overall survival (OS). The data will be analyzed for DFS and OS according to the BMI subgroups as well as two treatment arms (tamoxifen v AIs). The frequency of adverse events will be used to assess safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal patients with breast cancer who have hormones receptor positive tumour as defined by the expression of oestrogen receptor (ER) and/or progesterone receptor (PR).
* patients with a tumour stage IB, IC, or II irrespective of nodal stage (< 10 positive nodes)

Exclusion Criteria:

* premenopausal patients,
* ER/PR negative

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-01 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From date of random assignment to the first event during 5 years
  Event in the form of locoregional recurrence, distant metastasis, cancer in the contralateral breast, second primary cancer, or death from any cause.

SECONDARY OUTCOMES:
recurrence-free survival . | From date of randomization until the date of first documented progression during 5 years
  Disease specific mortality
overall survival (OS) | From day of diagnosis till date of death from disease/ other cause over an average of 5 years
  Till death due to disease/ other cause over an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Budhi S Yadav, MD, Principal Investigator — Post Graduate Institute of Medical Education & Research, Chandigarh, India
Locations (1):
- Department of Radiotherapy, Post Graduate Institute of Medical Education & Research, Chandigarh, India